CLINICAL TRIAL: NCT07366086
Title: Multicenter, Safety Follow-up Study to Assess Safety of Prior Treatment With Romosozumab in Children and Adolescents With Osteogenesis Imperfecta
Brief Title: Pediatric Safety Follow-up Study of Prior Treatment With Romosozumab for Osteogenesis Imperfecta
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220043; 2023-503293-21-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: Romosozumab; EVENITY
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of Care (Other): Participants who completed romosozumab trial 20200105 will continue to receive standard of care treatment (calcium and vitamin D), as determined by the investigator and local guidance. No investigational drug product will be administered in this trial as this is a safety follow-up.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants are recommended to receive Vitamin D supplements as standard of care treatment, per investigator discretion and local guidance.
Dietary Supplement: Calcium — Participants are recommended to receive Calcium supplements as standard of care treatment, per investigator discretion and local guidance.

SUMMARY:
The primary objective of this trial is to evaluate the safety of romosozumab in participants with osteogenesis imperfecta (OI) that have completed Study 20200105, regardless of whether they received investigational product (romosozumab) until the last protocol-specified dose or ended investigational product early.

ELIGIBILITY:
Inclusion Criteria:

- Participant has provided informed consent/assent prior to initiation of any trial specific activities/procedures.

OR Participant's legally authorized representative has provided informed consent when the participant is legally too young to provide informed consent, and the participant has provided written assent based on local regulations and/or guidelines prior to any trial-specific activities/procedures being initiated.

- Participant was randomized to the romosozumab arm and completed Trial 20200105 through the Month 15 Visit, regardless of whether they received investigational product (romosozumab) until the last protocol-specified dose or ended investigational product early.

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug trial, or less than 2 years since ending treatment on another investigational device or drug trial(ies) with the exception of trial 20200105. Other investigational procedures while participating in this trial are excluded.
* Participant likely to not be available to complete all protocol-required trial visits or procedures, and/or to comply with all required trial procedures to the best of the participant and investigator's knowledge.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Estimated)
Dates: Start 2026-03-07 (Estimated); Primary Completion 2028-05-21 (Estimated); Study Completion 2028-05-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com